CLINICAL TRIAL: NCT00127621
Title: Early Tracheotomy Versus Prolonged Endotracheal Intubation in Intensive Care Unit Patients
Brief Title: Early Tracheotomy Versus Prolonged Endotracheal Intubation in Intensive Care Unit (ICU) Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRACHEO
Record Dates: First submitted 2005-08-05; First posted 2005-08-08 (Estimated); Last update posted 2005-08-25 (Estimated); Status verified 2005-08

CONDITIONS: Respiratory Insufficiency
Keywords: ICU patients needing prolonged ventilatory support
MeSH Terms: conditions — Respiratory Insufficiency

INTERVENTIONS:
Procedure: early tracheotomy
Procedure: prolonged endotracheal intubation

SUMMARY:
This is a phase III trial comparing early tracheotomy versus prolonged endotracheal intubation in intensive care unit patients needing prolonged ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* Patients under ventilation support for at least 4 days
* Patients needing ventilatory support for > 7 days
* Age > 18 years
* Informed consent signed

Exclusion Criteria:

* Patients previously tracheotomised
* Major hemorrhagic risk
* Patients previously randomised in a trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468
Dates: Start 2002-04; Study Completion 2005-04

PRIMARY OUTCOMES:
28 days mortality
cumulated incidence of nosocomial pneumonia between days 1 and 28
number of ventilatory free days between days 1 and 28

SECONDARY OUTCOMES:
time in the ICU
time on mechanical ventilation
60 days mortality
number of septic episodes
accidental extubation
amount of sedation

CONTACTS AND LOCATIONS:
Overall Officials: François BLOT, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France